CLINICAL TRIAL: NCT00395382
Title: Randomised Controlled Trial of the Effect of Alendronate on Vascular Calcification and Arterial Stiffness in Chronic Kidney Disease: A Pilot Study
Brief Title: Study of the Effect of Alendronate on Vascular Calcification and Arterial Stiffness in Chronic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Monash University (Other)
Responsible Party: Dr Nigel Toussaint, Department of Nephrology, Monash Medical Centre, Clayton, Australia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HREC 06099C
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Vascular Calcification; Arteriosclerosis
Keywords: Vascular calcification; Arterial stiffness; Cardiovascular risk; Bone mineral metabolism; Calcium
MeSH Terms: conditions — Vascular Calcification; Arteriosclerosis | interventions — Alendronate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Alendronate
  Interventions: Drug: Alendronate
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alendronate — 70mg weekly orally
  Other Names: Fosamax
  Arms: 1
Drug: Placebo — weekly orally
  Arms: 2

SUMMARY:
Cardiovascular disease (CVD) is the commonest cause of mortality in patients with chronic kidney disease (CKD) and end-stage kidney disease (ESKD). Reasons for the greater incidence of CVD in this group include traditional CVD risk factors of hypertension, dyslipidemia and diabetes but more importantly also include non-traditional risk factors such as calcium and phosphate imbalance. The latter is thought most likely to contribute to vascular calcification, especially for those on dialysis, and this in turn leads to arterial stiffness and left ventricular hypertrophy, the two commonest cardiovascular complications. Arterial stiffness and calcification have been found to be independent predictors of all-cause and cardiovascular mortality in CKD. Few studies, though, have looked at both structural and functional changes associated with calcification and there have been very few interventional studies addressing this issue.

Control of calcium and phosphate levels in CKD can occur with the use of medications that reduce elevated serum phosphate (phosphate binders, mostly calcium-based) and those to treat hyperparathyroidism (vitamin D and more recently calcium sensing receptor agonists called calcimimetics). These pharmacological managements addressing calcium and phosphate imbalance reduce vascular calcification and CVD. Bisphosphonate therapy may also have a role in reduction of calcification.

Low bone mineral density (BMD) is common in CKD patients and predicts increased fracture risk similar to the general population. Bisphosphonate therapy improves BMD and lowers the fracture risk. Bisphosphonates may also have a role in secondary hyperparathyroidism to reduce hypercalcemia and allow for more aggressive calcitriol treatment. Recent studies have addressed the possibility of bisphosphonates reducing the progression of vascular calcification in CKD and revealed that the extent of calcification may be suppressed in association with a reduction in chronic inflammatory responses.

The investigators aim to perform a prospective, randomised study assessing the impact of alendronate on cardiovascular and bone mineral parameters. This will be a single-centre study involving subjects with CKD Stage 3 (those patients with GFR between 30 and 59ml/min). Arterial stiffness (by pulse wave analysis and pulse wave velocity) and vascular calcification (using CT scans through superficial femoral artery) will be followed as well as serum markers of calcium, phosphate and PTH. Differences in these end-points will be compared between participants taking alendronate and those not. The study will be conducted over a 12 month period and the investigators aim to recruit about 50 patients (25 on alendronate and 25 control).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with CKD Stage 3 (GFR between 30 and 59ml/min)
* Subjects must be 18 years of age or older
* Willingness to provide written informed consent

Exclusion Criteria:

* Subjects unable to give informed consent or whom have an expected life-span of less than 3 months
* Subjects undertaking renal replacement therapy (dialysis or transplantation)
* Subjects already taking bisphosphonates
* Subjects with recent fracture (within the last 3 months)
* Subjects scheduled to have a kidney transplant from a known living donor
* Subjects with active gastro-oesophageal reflux disease or peptic ulcer disease
* Subjects who are pregnant or planning on becoming pregnant in the next 18 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change in degree of arterial stiffness measured by pulse wave velocity | 18 months
Changes in vascular calcification on CT scans of superficial femoral artery and aorta | 18 months

SECONDARY OUTCOMES:
Changes in bone mineral density | 18 months
Changes in serum calcium and phosphate levels | 18 months
Cardiovascular events including myocardial ischaemia, myocardial infarction, cardiac failure, stroke, PVD | 18 months
Incidence of fractures | 18 months
Symptoms and severity of side effects from alendronate | 18 months
Episodes of hypocalcemia (serum corrected calcium <2.10mmol/L) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter G Kerr, MBBS FRACP, Principal Investigator — Monash Medical Centre, Clayton, Victoria, Australia
Locations (1):
- Department of Nephrology, Monash Medical Centre, Clayton, Victoria, Australia

REFERENCES:
- [Derived] Hara T, Hijikata Y, Matsubara Y, Watanabe N. Pharmacological interventions versus placebo, no treatment or usual care for osteoporosis in people with chronic kidney disease stages 3-5D. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013424. doi: 10.1002/14651858.CD013424.pub2. PMID 34231877
- [Derived] Toussaint ND, Lau KK, Strauss BJ, Polkinghorne KR, Kerr PG. Using vertebral bone densitometry to determine aortic calcification in patients with chronic kidney disease. Nephrology (Carlton). 2010 Aug;15(5):575-83. doi: 10.1111/j.1440-1797.2010.01288.x. PMID 20649879